CLINICAL TRIAL: NCT04087720
Title: A Multicenter, Open-Label, Efficacy and Safety Study of Pegloticase in Patients With Uncontrolled Gout Who Have Undergone Kidney Transplantation
Brief Title: Study of Pegloticase in Participants With Uncontrolled Gout Who Have Had a Kidney Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-KRY-406
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Uncontrolled Gout; Kidney Transplant
MeSH Terms: interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegloticase (Experimental): Participants receive 8 mg pegloticase every 2 weeks from Day 1 through Week 22
  Interventions: Biological: Pegloticase

INTERVENTIONS:
Biological: Pegloticase — intravenous (IV) infusion

SUMMARY:
The primary objective of this study is to evaluate the effect of pegloticase on the response rate of sustained serum uric acid (sUA) reduction to sUA < 6 mg/dL during Month 6 of treatment.

DETAILED DESCRIPTION:
The study design includes: 1) a Screening Period, lasting up to 35 days; 2) a 24-week treatment period which includes an End-of-Study (Week 24) /Early Termination Visit; 3) a safety follow-up phone/email Visit 30 days after the last infusion; and 4) a 3 month post-treatment follow up visit.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent;
* Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study;
* Adult men or women ≥ 18 years of age;
* Is a recipient of a de novo kidney from a living or deceased donor and is >1 year post transplant prior to screening;
* Is on a stable standard of care immunosuppression therapy for at least 3 months prior to screening;
* Kidney allograft is functional at entry, based on an estimated glomerular filtration rate (eGFR) ≥ 15 mL/min/1.73m²;
* Women of childbearing potential have a negative screening serum pregnancy test and will be required to use a medically approved form of birth control during their participation in the study;
* Uncontrolled gout, defined as:

  1. Hyperuricemia during screening as documented by sUA ≥ 7 mg/dL during Screening and prior to entry into the Treatment Period (Note: the sUA may be repeated up to 3 times during the Screening Period to confirm eligibility), and
  2. Inability to maintain sUA <6 mg/dL on other urate-lowering therapy or intolerable side effects or contraindicated with conventional urate-lowering therapy, and
  3. At least 1 of the following:

  i. Evidence of tophaceous deposits; ii. Recurrent gout flares defined as 2 or more flares in the 12 months prior to Screening; iii. Presence of chronic gouty arthritis;
* Able to tolerate low-dose prednisone (< 10 mg/day) as part of the required standard gout flare prophylaxis regimen for ≥ 1 week before the first infusion.

Exclusion Criteria:

* Any other organ transplant beside kidney;
* Any severe infection, unless treated and completely resolved at least 2 weeks prior to Day 1;
* Chronic or active hepatitis B virus infection;
* Known history of hepatitis C virus ribonucleic acid (RNA) positivity unless treated and viral load is negative;
* Known history of human immunodeficiency virus (HIV) positivity;
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency (tested at the Screening Visit);
* Decompensated congestive heart failure or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or uncontrolled blood pressure (> 160/100 mm Hg) at the end of the Screening Period (Day 1 prior to infusion);
* Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner, or not using an effective form of birth control, as determined by the Investigator;
* Prior treatment with pegloticase, another recombinant uricase (rasburicase), or concomitant therapy with a polyethylene glycol-conjugated drug;
* Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product;
* Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1, or plans to take an investigational drug during the study;
* Currently receiving systemic or radiologic treatment for ongoing cancer;
* History of malignancy within 5 years other than non-melanoma skin cancer, in situ carcinoma of cervix, early stage renal cell cancer or early stage prostate cancer that has been completely resected > 2 years prior to screening;
* Uncontrolled hyperglycemia with a plasma glucose value > 240 mg/dL at Screening that is not subsequently controlled by the end of the Screening Period;
* Diagnosis of osteomyelitis;
* Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome;
* Unsuitable candidate for the study, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the study;
* Currently receiving allopurinol, febuxostat or other urate lowering medications and unable to discontinue medication 7 days prior to Day 1; or
* Currently receiving probenecid and unable to discontinue medication within 3 days, prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (8):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Nephrology Consultants, Huntsville, Alabama
  - Keck School of Medicine of USC, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Genesis Clinical Research, Tampa, Florida
  - Coastal Medical Research, Brunswick, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Clear Lake Specialties, Webster, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Dalbeth N, Abdellatif A, Botson JK, Saag KG, Kumar A, Padnick-Silver L, Vranic Z, Marder BA, Becce F. Monosodium Urate Crystal Depletion and Bone Erosion Response in Kidney Transplant Recipients With Uncontrolled Gout Treated With Pegloticase: PROTECT Serial Dual-Energy Computed Tomography Findings. Transplant Direct. 2025 May 12;11(6):e1803. doi: 10.1097/TXD.0000000000001803. eCollection 2025 Jun. PMID 40371056
- [Derived] Abdellatif A, Zhao L, Chamberlain J, Cherny K, Xin Y, Marder BA, Scandling JD, Saag K. Pegloticase efficacy and safety in kidney transplant recipients; results of the phase IV, open-label PROTECT clinical trial. Clin Transplant. 2023 Sep;37(9):e14993. doi: 10.1111/ctr.14993. Epub 2023 May 3. PMID 37138473

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegloticase: Participants received 8 mg pegloticase by intravenous (IV) infusion every 2 weeks from Day 1 through Week 22
Period: Overall Study
Arm/Group | Pegloticase
Started | 20
Completed | 15
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawal by Subject - COVID-19 Concerns | 3

BASELINE CHARACTERISTICS:
Groups:
- Pegloticase: Participants received 8 mg pegloticase by IV infusion every 2 weeks from Day 1 through Week 22
Arm/Group | Pegloticase
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 9
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Serum Uric Acid (sUA) < 6 mg/dL Responders During Month 6
Description: sUA < 6 mg/dL responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 6, which includes pre-infusion and post-infusion results at Week 20, results at Week 21, pre-infusion and post-infusion results at Week 22, results at Week 23, results at Week 24, and unscheduled assessments of sUA collected between Week 20 and Week 24. Two-sided Exact Clopper-Pearson confidence interval is used for the calculation of the 95% confidence interval.
Time Frame: Month 6 (Weeks 20, 21, 22, 23, 24)
Population: Intent-to-treat (ITT) population: participants who received at least 1 dose of pegloticase. Participants in the ITT population with no lapse or cessation in treatment due to COVID-19 prior to the analysis time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 18
percentage of participants | 88.9 [65.3 to 98.6]

2. Secondary Outcome: Percentage of sUA < 5 mg/dL Responders During Month 6
Description: sUA < 5 mg/dL responders are defined as participants achieving and maintaining sUA <5 mg/dL for at least 80% of the time during Month 6, which includes pre-infusion and post-infusion results at Week 20, results at Week 21, pre-infusion and post-infusion results at Week 22, results at Week 23, results at Week 24, and unscheduled assessments of sUA collected between Week 20 and Week 24. Two-sided Exact Clopper-Pearson confidence interval is used for the calculation of the 95% confidence interval.
Time Frame: Month 6 (Weeks 20, 21, 22, 23, and 24)
Population: ITT population: participants who received at least 1 dose of pegloticase. Participants in the ITT population with no lapse or cessation in treatment due to COVID-19 prior to the analysis time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 18
percentage of participants | 88.9 [65.3 to 98.6]

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Pain Visual Analog Scale (VAS) Score Through Week 24
Description: The HAQ-Pain score consists of a doubly anchored, horizontal VAS 15 cm in length, and rates a participant's pain over the past week from 0 to 100 with 0 = no pain and 100 = severe pain. Baseline is defined as the last measurement taken prior to the first infusion of pegloticase. The 95% confidence interval is a two-sided normal theory-based 95% confidence interval.
Time Frame: Baseline, Weeks 6, 14, 20, 24
Population: ITT population: participants who received at least 1 dose of pegloticase. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegloticase
Number analyzed (Participants) | 20
score on a scale
  Change at Week 6: number analyzed (Participants) | 19
  Change at Week 6 | -16.11 (29.230)
  Change at Week 14: number analyzed (Participants) | 18
  Change at Week 14 | -34.81 (24.025)
  Change at Week 20: number analyzed (Participants) | 17
  Change at Week 20 | -34.63 (27.543)
  Change at Week 24: number analyzed (Participants) | 14
  Change at Week 24 | -33.05 (31.590)

4. Secondary Outcome: Change From Baseline in Heath Assessment Questionnaire - Disability Index (HAQ-DI) Score Through Week 24
Description: The HAQ-DI is a self-reported assessment of how a participant's illness affects their ability to function in their daily life over the past week. The HAQ-DI for a participant is calculated as the mean of the following 8 category scores: Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities. The HAQ-DI ranges from 0 to 3 with higher values indicating higher disability. Baseline is defined as the last measurement taken prior to the first infusion of pegloticase. The 95% confidence interval is a two-sided normal theory-based 95% confidence interval.
Time Frame: Baseline, Weeks 6, 14, 20, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegloticase
Number analyzed (Participants) | 20
score on a scale
  Change at Week 6: number analyzed (Participants) | 19
  Change at Week 6 | -0.30 (0.522)
  Change at Week 14: number analyzed (Participants) | 18
  Change at Week 14 | -0.52 (0.616)
  Change at Week 20: number analyzed (Participants) | 18
  Change at Week 20 | -0.38 (0.523)
  Change at Week 24: number analyzed (Participants) | 15
  Change at Week 24 | -0.25 (0.611)

ADVERSE EVENTS:
Time Frame: From the date of first dose of treatment through 30 days after the last dose of treatment (up to Week 22 plus 30 days).
Arm/Group | Pegloticase
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegloticase (N=20)
Atrial fibrillation (Cardiac disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Enterocolonic fistula (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegloticase (N=20)
Tachycardia (Cardiac disorders) | 1
Inner ear disorder (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 2
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT04087720/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT04087720/SAP_001.pdf